CLINICAL TRIAL: NCT06355882
Title: Cardiovascular Events in Patients With Low Cardiac Output Undergoing Local Dental Anesthesia With and Without Epinephrine: Randomized, Double-blind Pilot Study
Brief Title: Patients With Low Cardiac Output Syndrome Undergoing Local Dental Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Itamara Lucia Itagiba Neves, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCOSDental
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Low Cardiac Output Syndrome
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grupo de estudo (Lidocaine with epinephrine) (Active Comparator): Anesthetic lidocaine 2% with epinephrine 1:100.000
  Interventions: Procedure: Anesthetic infiltration
- Grupo controle (Lidocaine) (Active Comparator): Anesthetic lidocaine 2%
  Interventions: Procedure: Anesthetic infiltration

INTERVENTIONS:
Procedure: Anesthetic infiltration — Application of local dental anesthesia with two cartridges (3,6 mL) for dental procedures (tooth extraction or periodontal treatment) in patients with low cardiac output syndrome.

SUMMARY:
Patients with low cardiac output syndrome requiring surgical and periodontal dental treatment will be selected to undergo the dental procedure using local dental anesthetic: 2% lidocaine with epinephrine and 2% lidocaine without vasoconstrictor. Cardiovascular events and the safety of using two cartridges (3.6 mL) will be evaluated. They will be evaluated by Holter monitoring in the period of 1 hour before, during and 1 hour after the procedure and blood pressure correction will be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced heart failure, in INTERMACS III using dobutamine at 5 to 20 µg/kg/minute due to low cardiac output syndrome
* Presence of periodontal disease, in the 4th or 6th sextant with indication of supragingival and/or subgingival periodontal scaling;
* Residual root or teeth with periodontal disease in the jaw, with simple extraction indicated.

Exclusion Criteria:

* Patients with a ventricular assist device such as an intra-aortic balloon implanted less than 24 hours after the dental procedure or with extracorporeal membrane oxygenation (ECMO);
* Using other inotropes;
* On mechanical ventilation;
* Continuously using a non-invasive ventilation mask;
* In septic shock;
* Presence of acute myocardial infarction <30 days;
* Patients with terminal non-cardiac disease, cyanotic congenital heart disease or cardiomyopathies with arrhythmogenic potential (arrhythmogenic dysplasia, hypertrophic cardiomyopathy, non-compacted myocardium);
* Pregnant women;
* History of sudden death recovered < 1 month ago;
* In the recent postoperative period of cardiac surgery (5 days);
* Allergic to sodium bisulfite and methylparaben, preservatives of epinephrine and the anesthetic cartridge, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Amount ventricular and supraventricular arrhythmia | during dental procedures
  Number of ventricular and supraventricular arrhythmias recorded using Holter

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After thesis defense, the IPD will be available on the Portal Digital Library of Theses and Dissertations of the University of São Paulo (http://www.teses.usp.br/index.php?option=com_jumi&fileid=12&Itemid=77&lang=pt-br), in a PDF file.
Supporting Information: CSR

REFERENCES:
- [Background] Comite Coordenador da Diretriz de Insuficiencia Cardiaca; Rohde LEP, Montera MW, Bocchi EA, Clausell NO, Albuquerque DC, Rassi S, Colafranceschi AS, Freitas AF Junior, Ferraz AS, Biolo A, Barretto ACP, Ribeiro ALP, Polanczyk CA, Gualandro DM, Almeida DR, Silva ERR, Figueiredo EL, Mesquita ET, Marcondes-Braga FG, Cruz FDD, Ramires FJA, Atik FA, Bacal F, Souza GEC, Almeida GLG Junior, Ribeiro GCA, Villacorta H Junior, Vieira JL, Souza JD Neto, Rossi JM Neto, Figueiredo JA Neto, Moura LAZ, Goldraich LA, Beck-da-Silva L, Danzmann LC, Canesin MF, Bittencourt MI, Garcia MI, Bonatto MG, Simoes MV, Moreira MCV, Silva MMF, Olivera MT Junior, Silvestre OM, Schwartzmann PV, Bestetti RB, Rocha RM, Simoes R, Pereira SB, Mangini S, Alves SMM, Ferreira SMA, Issa VS, Barzilai VS, Martins WA. Diretriz Brasileira de Insuficiencia Cardiaca Cronica e Aguda. Arq Bras Cardiol. 2018 Sep;111(3):436-539. doi: 10.5935/abc.20180190. No abstract available. Portuguese. PMID 30379264
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW. 2009 focused update incorporated into the ACC/AHA 2005 Guidelines for the Diagnosis and Management of Heart Failure in Adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the International Society for Heart and Lung Transplantation. Circulation. 2009 Apr 14;119(14):e391-479. doi: 10.1161/CIRCULATIONAHA.109.192065. Epub 2009 Mar 26. No abstract available. PMID 19324966
- [Background] Bacal F, Marcondes-Braga FG, Rohde LEP, Xavier Junior JL, Brito FS, Moura LAZ, Colafranceschi AS, Lavagnoli CFR, Gelape CL, Almeida DR, Gaiotto FA, Atik FA, Figueira FAMS, Souza GEC, Rodrigues H, Campos IW, Souza Neto JD, Rossi Neto JM, Gasparetto J, Goldraich LA, Benvenuti LA, Seguro LFBC, Ulhoa Junior MB, Moreira MDCV, Avila MS, Carneiro R, Mangini S, Ferreira SMA, Strabelli TM. 3 feminine Diretriz Brasileira de Transplante Cardiaco. Arq Bras Cardiol. 2018 Aug;111(2):230-289. doi: 10.5935/abc.20180153. No abstract available. Portuguese. PMID 30335870
- [Background] Oliveira ACG, Neves ILI, Sacilotto L, Olivetti NQS, Santos-Paul MAD, Montano TCP, Carvalho CMA, Wu TC, Grupi CJ, Barbosa SA, Pastore CA, Samesima N, Hachul DT, Scanavacca MI, Neves RS, Darrieux FCC. Is It Safe for Patients With Cardiac Channelopathies to Undergo Routine Dental Care? Experience From a Single-Center Study. J Am Heart Assoc. 2019 Aug 6;8(15):e012361. doi: 10.1161/JAHA.119.012361. Epub 2019 Jul 19. PMID 31319747
- [Background] Laragnoit AB, Neves RS, Neves IL, Vieira JE. Locoregional anesthesia for dental treatment in cardiac patients: a comparative study of 2% plain lidocaine and 2% lidocaine with epinephrine (1:100,000). Clinics (Sao Paulo). 2009;64(3):177-82. doi: 10.1590/s1807-59322009000300005. PMID 19330241
- [Background] Neves IL, Avila WS, Neves RS, Giorgi DM, Santos JF, Oliveira Filho RM, Grupi CJ, Grinberg M, Ramires JA. Maternal-fetal monitoring during dental procedure in patients with heart valve disease. Arq Bras Cardiol. 2009 Nov;93(5):463-742. doi: 10.1590/s0066-782x2009001100005. PMID 20084307
- [Background] Neves RS, Neves IL, Giorgi DM, Grupi CJ, Cesar LA, Hueb W, Grinberg M. Effects of epinephrine in local dental anesthesia in patients with coronary artery disease. Arq Bras Cardiol. 2007 May;88(5):545-51. doi: 10.1590/s0066-782x2007000500008. English, Portuguese. PMID 17589629
- [Background] Ruffolo RR Jr. The pharmacology of dobutamine. Am J Med Sci. 1987 Oct;294(4):244-8. doi: 10.1097/00000441-198710000-00005. PMID 3310640
- [Background] Leier CV, Webel J, Bush CA. The cardiovascular effects of the continuous infusion of dobutamine in patients with severe cardiac failure. Circulation. 1977 Sep;56(3):468-72. doi: 10.1161/01.cir.56.3.468. PMID 884803
- [Background] Jewitt D, Birkhead J, Mitchell A, Dollery C. Clinical cardiovascular pharmacology of dobutamine. A selective inotropic catecholamine. Lancet. 1974 Aug 17;2(7877):363-7. doi: 10.1016/s0140-6736(74)91754-1. No abstract available. PMID 4136593
- [Background] Tuttle RR, Mills J. Dobutamine: development of a new catecholamine to selectively increase cardiac contractility. Circ Res. 1975 Jan;36(1):185-96. doi: 10.1161/01.res.36.1.185. PMID 234805
- [Background] Binner C, Wagner J, Schmalz G, Eisner M, Rast J, Kottmann T, Haak R, Oberbach A, Borger MA, Garbade J, Ziebolz D. Insufficient Oral Behaviour and the High Need for Periodontal Treatment in Patients with Heart Insufficiency and after Heart Transplantation: A Need for Special Care Programs? J Clin Med. 2019 Oct 12;8(10):1668. doi: 10.3390/jcm8101668. PMID 31614807
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Dajani AS, Taubert KA, Wilson W, Bolger AF, Bayer A, Ferrieri P, Gewitz MH, Shulman ST, Nouri S, Newburger JW, Hutto C, Pallasch TJ, Gage TW, Levison ME, Peter G, Zuccaro G Jr. Prevention of bacterial endocarditis: recommendations by the American Heart Association. J Am Dent Assoc. 1997 Aug;128(8):1142-51. doi: 10.14219/jada.archive.1997.0375. PMID 9260427